CLINICAL TRIAL: NCT01905124
Title: A Phase 2, Randomized, Double-Masked, Placebo-Controlled Study of the Safety and Efficacy of Daily CF101 Administered Orally to Subjects With Active, Sight-Threatening, Noninfectious Intermediate or Posterior Uveitis
Brief Title: Safety &Efficacy of CF101 to Subjects With Uveitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The company has decided not to conduct the study
Sponsor: Can-Fite BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CF101-241UV
Record Dates: First submitted 2013-07-14; First posted 2013-07-23 (Estimated); Last update posted 2018-02-01 (Actual); Status verified 2018-01

CONDITIONS: Uveitis, Posterior; Uveitis, Intermediate
Keywords: Uveitis; Intermediate uveitis; Posterior uveitis
MeSH Terms: conditions — Uveitis, Posterior; Uveitis, Intermediate; Uveitis | interventions — CF101; N(6)-(3-iodobenzyl)-5'-N-methylcarboxamidoadenosine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Drug: CF101 (Experimental): CF101 1 mg q12 hours
  Interventions: Drug: CF101
- Placebo tablets of CF101 (Placebo Comparator): Placebo tablets q12 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CF101 — CF101 1 mg tablets orally every 12 hours for 24 weeks
  Other Names: IB-MECA
  Arms: Drug: CF101
Drug: Placebo — Matching placebo tablets orally every 12 hours for 24 weeks
  Other Names: Sugar pills
  Arms: Placebo tablets of CF101

SUMMARY:
This is a Phase 2, randomized, double-masked, placebo-controlled study subjects with active, sight-threatening, noninfectious intermediate or posterior uveitis.

DETAILED DESCRIPTION:
This is a Phase 2, randomized, double-masked, placebo-controlled study in adult males and females, aged 18 years and over, with active, sight-threatening, noninfectious intermediate or posterior uveitis. Subjects will be randomly assigned to receive CF101 1 mg or matching placebo tablets in a 2:1 ratio orally every 12 hours for 24 weeks.

At the Screening Visit (performed within 4 weeks prior to Baseline), subjects who provide written informed consent will have a complete medical history, medication history, physical examination, weight, sitting blood pressure, pulse rate, temperature, electrocardiogram (ECG), clinical laboratory tests, and ophthalmologic examination, including biomicroscopy and grading of uveitis activity. For assessment of uveitis activity and response to treatment, fundus photography will be obtained according to a standardized procedure and interpreted at the Uveitis Photograph Reading Center.

Subjects who successfully qualify will begin dosing with CF101 1 mg or placebo, to be taken orally every 12 hours for 24 weeks. At the Baseline Visit, a PBMC sample will be obtained for assessment of A3AR expression level. Subjects will return for safety and efficacy assessments and a new supply of study medication at Weeks 2, 4, 8, 12, 16, 20, and for final assessment and discharge at Week 24. A telephone call to each subject will be made at Week 26, for the purpose of collecting information on adverse events (AEs) and concomitant medications.

During the course of the trial, concomitant use of intraocular or posterior subtenon corticosteroids, intravitreal injections (including but not limited to steroids or anti-vascular endothelial growth factors), systemic corticosteroids at a dose >20 mg/day prednisone equivalent, or monoclonal antibody therapy is prohibited. Systemic corticosteroid and immunosuppressive regimens must remain stable throughout the course of the trial.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years of age and over;
2. Diagnosis of active, sight-threatening, noninfectious intermediate or posterior uveitis, as determined by the Standardization of Uveitis Nomenclature (SUN) Working Group Criteria.
3. Vitreous haze in at least 1 eye (the "study eye") of ≥Grade 3 on the "Miami Scale" at the Screening Visit, as confirmed by the Uveitis Photograph Reading Center; ,
4. Best corrected visual acuity (BCVA) in the poorer seeing eye of 1.3 logarithm of the minimum angle of resolution (logMAR) or better by Early Treatment Diabetic Retinopathy Study (ETDRS; equivalent to 20/400) at Screening;
5. Requires, in the judgment of the Investigator, systemic therapy to treat uveitis;
6. No plans for elective ocular surgery during the trial duration;

10. Ability to understand and provide written informed consent.

Exclusion Criteria:

1. Primary diagnosis of anterior uveitis;
2. Uveitis of infectious etiology;
3. Presence of chorioretinal scars that are highly suspicious for ocular toxoplasmosis;
4. Confirmed or suspected uveitis of traumatic etiology;
5. Clinically suspected or confirmed central nervous system or ocular lymphoma;
6. Presence of any other form of ocular malignancy in the either eye including choroidal melanoma;
7. Corneal or lens opacities or obscured ocular media other than vitreous haze upon enrollment such that reliable clinical evaluations and grading of the posterior segment cannot be performed;
8. Pupillary dilation inadequate for quality fundus photography;
9. Uncontrolled glaucoma or ocular hypertension in either eye, defined as intraocular pressure (IOP) >21 mm Hg while on medical therapy;
10. Chronic hypotony (IOP <6 mm Hg) in either eye;
11. Presence of an ocular implantable steroid-eluting device;
12. Ocular injection of corticosteroid within 3 months prior to Baseline;
13. Use of Retisert within 6 months prior to baseline;
14. Use of the following within 90 days prior to Baseline or anticipated use to either eye during the trial:

    1. Intravitreal injections (including but not limited to steroids or anti-vascular endothelial growth factors), or
    2. Posterior subtenon steroids;
15. YAG capsulotomy within 30 days prior to Day 1 in the study eye;
16. History of herpetic infection in the study eye or adnexa;
17. Oral corticosteroid dose >20 mg/day prednisone equivalent;
18. Oral corticosteroid dose has been changed within 2 weeks prior to screening, or is expected to change while on study;
19. Systemic immunosuppressive agent dose has been changed within 2 weeks prior to screening;
20. Treatment with systemic monoclonal antibody within the longer of 1 month or 5 serum half-lives, prior to screening;
21. Diagnosis or history of Behçet's Disease;
22. Any significant ocular disease that could compromise vision in either eye, including but not limited to:

    1. Diabetic retinopathy: proliferative diabetic retinopathy or non-proliferative diabetic retinopathy that compromise vision,
    2. Wet age-related macular degeneration, and
    3. Myopic degeneration with active subfoveal choroidal neovascularization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2019-09 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Severity of uveitis on standardized photographic assessment | 24 weeks
  Standardized fundus photographs will be obtained and uniformly assessed in a masked fashion at the Reading Center

SECONDARY OUTCOMES:
Safety of CF101 | 24 weeks
  Frequency, nature, and severity of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Bnei-Zion Medical Center, Haifa, Israel